CLINICAL TRIAL: NCT04917458
Title: Effects of Cholecalciferol on Depressive Symptoms in Type 2 Diabetes Mellitus Patients: Study of Neurotrophin-3, Serotonin, and C-Peptide
Brief Title: Cholecalciferol on Depressive Symptoms in Type 2 Diabetes Mellitus Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr Rudi Putranto SpPD KPsi MPH, Lecturer, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-05-0484
Record Dates: First submitted 2021-04-21; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2; Depressive Symptoms
Keywords: Diabetes Mellitus, Type 2; Depression; Cholecalciferol
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression | interventions — Cholecalciferol; Capsules

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double blind, and controlled clinical study to investigate the effects of cholecalciferol on depressive symptoms in type 2 diabetes mellitus patients. Patients included into the study will be randomized into two groups and receive placebo (as control group) or cholecalciferol administered orally for 3 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients included into the study will be randomized into two groups and receive placebo (as control group) or 4000 IU Vitamin D (as therapy group) once a day for 90 days. Randomization and blinding code preparation will be performed by using block permuted randomization technique with a block size combination of 4 and 6. The randomized intervention code was hidden in a closed envelope to avoid knowing the sequence of the therapy given.
  All packaging and labeling of the study products will be prepared by Pharmacy Departement Ciptomangunkusumo General Hospital. The study products will be prepared in such packages which will be recognized as products for clinical trial only. In order to keep the blinding procedures, the study drugs will all be provided by Pharmacy Department in a double-blind double-dummy preparation. Placebo tablet will also be prepared by Pharmacy Department and made identical in appearance with the active tablets.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cholecalciferol (Experimental): -Vitamin D 25 (OH) 4000 IU capsules, tablet @ 1000 IU One capsule for once a day for 30 days of study period.
  Interventions: Drug: Cholecalciferol 4000 IU Oral Capsule, Liquid Filled
- Control Group (Placebo Comparator): Placebo will be administrated orally, One capsule once a day for 30 days of study period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol 4000 IU Oral Capsule, Liquid Filled — -Vitamin D 25 (OH) or Cholecalciferol 4000 IU capsules, each capsules contain Vitamin D3 tablet @ 1000 IU Patients included into the study will be randomized into two groups and receive placebo (as control group) or cholecalciferol administered orally for 3 months.
  Other Names: Vitamin D3
  Arms: Cholecalciferol
Drug: Placebo — Placebo will be given to control group. It would be administrated orally, one capsule once a day for 30 days of study period
  Arms: Control Group

SUMMARY:
One in eleven adults falls ill with Diabetes Mellitus (DM) and 90% of them suffered from type 2 DM. Depression in type 2 DM patients had a big impact, acting as a major barrier to self-care in type 2 DM patients. Depression in diabetes patients is also associated with decreasing quality of life. Poor self-care behavior and adherence, poor glycemic control, and increased risk of mortality about 36-38% from cardiovascular complications are other known debilitating results.

Vitamin D receptors are present in many organ systems, namely the pancreas, intestine, musculoskeletal, and nervous systems. Vitamin D has pleiotropic effects, which were seen from its mechanism as an anti-inflammatory, anti-apoptotic, and immunomodulatory agent. Based on the mechanism of Vitamin D action in the nervous system, which also plays a role in depression pathogenesis, vitamin D is hypothesized to have a beneficial effect on depression, both for depression prevention and treatment. Few studies denote that Vitamin D can improve depression in type 2 DM patients. Vitamin D may become an important adjuvant therapy to ameliorate depression in type 2 DM patients. These clinical trials concerning vitamin D in type 2 DM are relevant, reminding that type 2 DM resulted in higher morbidity, mortality, and numerous high-risk complications in the population.

DETAILED DESCRIPTION:
According to World Health Organization report's, depression was estimated causing distress in most people on 2030. 1 In Indonesia, the prevalence of depression in 2017 was 3,7%.2 Depression often found in Internal medicine patient's as a comorbid in various chronic diseases. 3 One of the most common chronic disease is type 2 diabetes mellitus. There's one in eleven adults suffered from diabetes mellitus, and 90% of them had type 2 diabetes mellitus (DM). Basic Health Research Data on 2018 showed there were 10.9% case type 2 DM in Indonesia. 4 DKI Jakarta Province had 3,4% or 11.226 people aged 15 years and over with Diabetes Mellitus and had been a highest prevalence of Diabetes Mellitus among population aged 15 years and over. Meanwhile, prevalence of depression among adults aged 15 and over in DKI Jakarta was 5.9%. Seminkovics K et al5 reported one in four people with type 2 diabetes mellitus suffered from depression in United States. In Indonesia, Nasrun WMS6 reported there were 27,6% prevalence of depression in type 2 diabetes mellitus patients's with cognitive impairment, while Arshita et al7 found there were 60% patients with depression in type 2 diabetes mellitus patients with pedic ulcers in RSCM .

Depression in type 2 Diabetes Mellitus patients had a big impact, such as: depression can be a major barrier to self-care in type 2 diabetes mellitus patients. 1,5 Depression in diabetes patients is also associated with decreasing quality of life. 6 Poor of self-care behavior and adherence, poor of glycemic control, and increased risk of mortality about 36-38% from cardiovascular complication are other known debilitating results. 8 Vitamin D receptors are present in various organs such as the pancreas, intestine, musculoskeletal, and nervous system. Vitamin D has a pleiotrophic effect which were seen from its mechanism as anti-inflammatory, anti-apoptotic, and immunomodulatory. 16 Based on mechanism of Vitamin D action in nervous system, which also plays a role in the depression pathogenesis, vitamin D is hypothesized to have a beneficial effect on depression, both for prevention and treat the pathomechanism. The protective effect of Vitamin D for prevent depression had been widely studied in copious observational epidemiological studies, although with diversified results. Many studies have been conducted to assess the beneficial effects of vitamin D on a variety outcomes including depression, which are summarized in systematic reviews and meta-analyzes of observational studies. A meta-analyses by Ju SY et al38 found that low plasma 25 (OH) D levels were associated with and increased risk of depression in a cross sectional study with 43,1377 participants.

Vitamin D deficiency is a worldwide health problem. Vitamin D had known as an important role in biological processes, calcium homeostasis, and various health problems. In addition to its role in musculoskeletal, vitamin D is also associated with a few non-musculoskeletal diseases such as immunity, cancer, cardiovascular disease, hypertension, diabetes, and psychological problems like dementia or depression. 17 Both Vitamin D and its analogues are natural ligands for vitamin D receptor (VDR). Vitamin D receptors are widely distributed throughout body including brain and pancreas. Vitamin D receptors found in cerebellum, hippocampus, substantia nigra, basal forebrain, prefrontal cortex and hypothalamus. This explains the role of vitamin D in brain development and emotional disorders. In brain development, vitamin D played role in proliferation and differentiation of neuron cells. In adult brain, vitamin D played a role in neurogenesis in the hippocampus and synthesizes neurotransmitters such as dopamine, GABA, and serotonin. 18 It's known as depression neurotransmitter.

Other studies showed that vitamin D might repair neurotransmitters, inflammation, metabolic, and oxidative stress. Cholecalciferol will activate 1-α hydroxylase enzymes and P450 cytochrome, which transformed calcifediol hydroxylation into activated vitamin D in central nervous system, so that improving depression. Anti depressants such as SSRIs (Selective serotonin reuptake inhibitors), can induce gastrointestinal bleeding in patients whose taking anti-platelets or anti-coagulants, increase weight and dyslipidemia. Thus, other studies therapy based on pathogenesis of depression, effective and side effects need to be done.

Few studies denote that Vitamin D can improve depression in type 2 DM patients. Those studies used only Beck Depression Inventory test to assess depression without any biological markers. Vitamin D may become an important adjuvant therapy to ameliorate depression in type 2 DM. These clinical trials concerning vitamin D in type 2 DM are relevant, reminding that type 2 DM resulted in higher morbidity, mortality and numerous high risk complication in the population.

Methods/Design: This is a prospective, randomized, double blind, and controlled clinical study to investigate the effects of cholecalciferol on depressive symptoms in type 2 diabetes mellitus patients. Patients included into the study will be randomized into two groups and receive placebo (as control group) or cholecalciferol administered orally for 3 months.

Discussion : Vitamin D may become an important adjuvant therapy to ameliorate depression in type 2 DM patients. Thus, type 2 diabetes mellitus with depression symptoms will have a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with aged 18 and over
* Living in around Jakarta
* Type 2 diabetes mellitus patients with depression symptom
* Patients with Body mass index 20-30 m/kg2
* Patients are able and willing to maintain diet, physical activity, and lifestyle for 3 months
* Patients are able and willing to control for follow up

Exclusion Criteria:

* - Presence of severe hepatic dysfunction, defined as cirrhosis hepatic
* Presence of severe renal dysfunction, defined as chronic kidney disease stage 5 or e-GFR ≤15 or history of hemodialysis
* Patients with acute coronary syndrome
* Presence of acute systemic inflammatory response syndrome (SIRS). The term SIRS describes a clinical state arising from a non-specific cause, infective, or otherwise
* Recent obtained vitamin D therapy within the last 3 months
* Current or regular use of corticosteroids within immunosuppressant dosage
* Presence of major depression
* Presence of psychosis
* Current or regular use of anti-depressant
* Current or regular use of phenytoin or phenobarbital
* For females: current pregnancy and lactation period
* Patients who refuse the studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Evaluating the effects of cholecalciferol for depression symptoms with BDI II score | 90 days
  Improvement rate on days 90 (end of study) as defined by a proportion of subjects with category of BDI II score below 13. The BDI II scale was a subjective measurement of depressive symptoms. Interpretation of BDI II were 0-13 for minimal depression, 14-19 for mild depression, 20-28 for moderate depression, and 29-63 for major depression. Cholecalciferol with doses of 4000 IU a day expected to demote BDI II scale or depressive symptoms in participants.

SECONDARY OUTCOMES:
Evaluating the effects of cholecalciferol against neuroplasticity (NT-3) | 30 days
  NT-3 concentration (pg/ml) in the sample was determined by comparing the sample against the standard curve. Some studies have shown that neurotrophin-3 (NT-3 pg/ml) levels decreased in depression. Thus, cholecalciferol (for doses of 4000 IU a day) with expected could increase NT-3 pg/ml plasm levels. Furthermore, the enhancement of NT-3 pg/ml concentrates expected to had correlated with scale BDI II improvement.
Evaluating the effects of cholecalciferol against serotonin | 30 days
  Studies have shown that serotonin (ng/mL) in depressive patients had lower levels than patient without depressive syndrome. The serotonin levels were measured by the ELISA method. Cholecalciferol expected could increase levels of serotonin concentration (ng/mL) significantly 2-3 times after administrated.
Evaluating the effects of cholecalciferol against C-Peptide | 30 days
  C-peptide hormone is an indicator of insulin secretion. Specifically, a c-peptide level of less than 0.2 nmol/l is associated with a diagnosis of type 1 diabetes mellitus. C-peptide measured using ELISA at a minimal room temperature for 24 hours. Cholecalciferol expected could improve C-peptide levels concentration in type 2 Diabetes Mellitus.

CONTACTS AND LOCATIONS:
Overall Officials: Rudi Putranto, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo National General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No